CLINICAL TRIAL: NCT00219336
Title: A Media Based Motivational Intervention to Reduce Alcohol Exposed Pregnancies (AEPs)
Brief Title: A Media Based Motivational Intervention to Prevent Alcohol Exposed Pregnancies (AEPs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda Sobell, Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U50/CCU300860; U50/CCU300860 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Alcohol Consumption; Fetal Alcohol Syndrome Disorders; Students
Keywords: Prevent Alcohol Exposed Pregnancies; Reduced Alcohol Used; Self-Guided Motivational Intervention; Effective Contraception; Contraception; College Students
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-motivational Choices (Experimental): Students and nonstudents were mailed a brochure prepared as part of the PHC study intervention, Making Healthy Choices for a Healthy Baby in English or Mujeres y Salud Eligiendo Opciones Saludables in Spanish. This brochure allows women to make informed decisions about preventing an AEP. The MF materials included nonstigmatizing messages about drinking and contraception embedded among other health messages. Similar to Project CHOICES, this group also received a brochure on birth control practices.
  Interventions: Behavioral: Self-guided Motivational Intervention
- Information Only (Active Comparator): Students and nonstudents were mailed a brochure prepared by the CDC. The brochure (English: Think Before You Drink: You Can Hurt Your Unborn Baby; Spanish: Piénselo Antes de Beber: Puede Lastimar a Su Futuro Bebe), available at the CDC website, targets women of childbearing-age, discusses FAS and the negative effects of a mother's drinking on her unborn child, and recommends calling Alcoholics Anonymous or an alcohol treatment program for help to stop drinking. The CDC brochure did not contain information about how to contracept effectively.
  Interventions: Behavioral: Informational Only

INTERVENTIONS:
Behavioral: Self-guided Motivational Intervention — Using a randomized two-group design, a self-guided motivational intervention based on Project CHOICES will be compared to an informational only intervention, both directed at preventing alcohol-exposed pregnancies (AEPs) with students and nonstudents. Participants will be women 18 to 44 years of age who are at risk of an AEP. All materials are sent to participants through the USPS.
  Arms: Self-motivational Choices
Behavioral: Informational Only — Using a randomized two-group design, an informational intervention using a brochure from the CDC will be compared to a self-guided motivational intervention based on Project CHOICES, both directed at preventing alcohol-exposed pregnancies (AEPs) with students and nonstudents. Participants will be women 18 to 44 years of age who are at risk of an AEP. All materials are sent to participants through the USPS
  Arms: Information Only

SUMMARY:
The study evaluated the effectiveness of a mail-based self-guided motivational intervention based on Project CHOICES to reduce alcohol-exposed pregnancies (AEP) with female students and non-students 18 to 44 years of age living in Florida. The investigators hypothesize that the motivational intervention will significantly reduce more women's risk of an AEP than will an informational intervention aimed at preventing fetal alcohol syndrome. Materials will be available in Spanish and English

DETAILED DESCRIPTION:
The proposed project will evaluate the effectiveness of a mail-based self-guided motivational intervention based on Project CHOICES to reduce alcohol-exposed pregnancies (AEP) among students and non-students. Participants will be women 18 to 44 years of age who are at risk of an AEP. The community targeted will be the state of Florida. Materials were available in Spanish and English The intervention will be based on the investigators' previous experience in (a) promoting self-change of drinking behavior at a community level and (b) preventing reduced risk for AEP through the use of a motivational interventional materials used in Project CHOICES. Using a 2 group randomized design, the self-guided motivational intervention will be compared to an intervention directed at preventing fetal alcohol syndrome (FAS). The FAS prevention condition, a brochure developed by the CDC, served as the standard treatment control group in that most information available at the community level concerning the effects of alcohol on the developing fetus relate to FAS (e.g., warning labels on alcoholic beverage containers). It is suggested that many women, particularly college students, at risk for AEP do not view themselves as at risk for FAS and therefore do not view FAS-oriented prevention messages as personally relevant. The proposed experimental design will evaluate a mail-based strategy that could be easily implemented throughout communities. The proposed study design will have more methodological rigor and allow a more careful evaluation than would be possible if the intervention was initially targeted at the entire community. The follow-up will be the entire 6-months post-intervention.If successful, this low-cost intervention can be readily disseminated throughout the local area. Specific objectives are as follows:

1. Develop an evidence-based intervention to reduce alcohol-exposed pregnancies that can be easily disseminated at a community level through the mail and other media outlets.
2. Implement the AEP prevention intervention using a randomized controlled trial with women recruited from a community at higher than normal risk for AEPs.
3. Evaluate the efficacy of the AEP prevention intervention for reducing AEP risk as compared to a community level intervention aimed at preventing FAS using the 3 primary outcome measures in previous Project CHOICES studies: (a) AEP reduced risk through reduced drinking or effective contraception, or both; (b) AEP reduced risk through drinking only; and (c) reduced risk through effective contraception only.
4. Disseminate results of the study to health care providers in the local community.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 44 years who are not pregnant, not trying to become pregnant, and able to bear children.
* At risk for an alcohol exposed pregnancy 90 days prior to the interview defined as:

  1. had heterosexual vaginal intercourse with ineffective contraception
  2. not effectively using contraception
  3. drinking either ≥ 8 drinks per week on average or ≥ 5 drinks in a single day or both
  4. returned their informed consent and assessment materials within 60 days after it was mailed to them

Exclusion Criteria:

* No alcohol consumption or vaginal intercourse in the 90 days prior to the interview
* Pregnant
* Trying to become pregnant
* Not able to bear children
* Using contraception effectively

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
AEP reduced risk through reduced drinking and effective contraception, or both | 6 months post intervention
  Not at risk if a women reported no risky drinking (see definition in outcome 2) or contracepting effectively, or both
AEP reduced risk through reduced drinking only | 6 months post intervention
  Reduced risk drinking defined as ≤ 7 standard drinks (SDs) per week and ≤ 4 SDs on any day during the 6-month follow-up interval; 1 SD = 14 g absolute alcohol.
AEP reduced risk through effective contraception only | 6 months post intervention
  The effectiveness of birth control methods was evaluated using algorithms (e.g., If you missed a pill during this time period, did you take both pills the next day and did you use a back up method other than rhythm or withdrawal until you started your next packet of pills?) from Project CHOICES

CONTACTS AND LOCATIONS:
Overall Officials: Linda C Sobell, Ph.D., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gioia CJ, Sobell LC, Sobell MB, Agrawal S. Craigslist versus print newspaper advertising for recruiting research participants for alcohol studies: Cost and participant characteristics. Addict Behav. 2016 Mar;54:24-32. doi: 10.1016/j.addbeh.2015.11.008. Epub 2015 Nov 19. PMID 26675247